CLINICAL TRIAL: NCT04998981
Title: A Phase 3, Multi-Center, Placebo- and Active-Controlled, Randomized, Double-Blind, 12-Week Study to Evaluate the Efficacy and Safety of K-877 in Chinese Patients With High TG and Low HDL-C
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of K-877 in Chinese Patients With High TG and Low HDL-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-877-3.01CH
Record Dates: First submitted 2021-07-14; First posted 2021-08-10 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Tablets; (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- K-877 0.1 mg BID (Experimental): K-877 0.1 mg tablet twice daily, Placebo tablet twice daily, Placebo capsule once daily
  Interventions: Drug: Placebo capsule; Drug: K-877 0.1 mg tablet; Drug: Placebo tablet
- K-877 0.2 mg BID (Experimental): K-877 0.1 mg tablet x 2 twice daily, Placebo capsule once daily
  Interventions: Drug: K-877 0.1 mg tablet; Drug: Placebo capsule
- Fenofibrate 200 mg QD (Active Comparator): Fenofibrate 200 mg capsule once daily, Placebo tablet x 2 twice daily
  Interventions: Drug: Fenofibrate 200 mg capsule; Drug: Placebo tablet
- Placebo (Placebo Comparator): Placcebo tablet x 2 twice daily, Placebo capsule once daily
  Interventions: Drug: Placebo tablet; Drug: Placebo capsule

INTERVENTIONS:
Drug: K-877 0.1 mg tablet — K-877 0.1 mg tablet x 2 twice daily
  Other Names: Pemafibrate
  Arms: K-877 0.2 mg BID
Drug: Fenofibrate 200 mg capsule — Fenofibrate 200 mg capsule once daily
  Arms: Fenofibrate 200 mg QD
Drug: Placebo tablet — Placebo tablet x 2 twice daily
  Other Names: Placebo tablet (matching K-877)
  Arms: Fenofibrate 200 mg QD; Placebo
Drug: Placebo capsule — Placebo capsule once daily
  Other Names: Placebo capsule (matching fenofibrate)
  Arms: K-877 0.1 mg BID; K-877 0.2 mg BID; Placebo
Drug: K-877 0.1 mg tablet — K-877 0.1 mg tablet twice daily
  Other Names: Pemafibrate
  Arms: K-877 0.1 mg BID
Drug: Placebo tablet — Placebo tablet twice daily
  Other Names: Placebo tablet (matching K-877)
  Arms: K-877 0.1 mg BID

SUMMARY:
A Phase 3 Study to Evaluate the Efficacy and Safety of K-877 in Chinese Patients with High TG and Low HDL-C

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all of the following criteria apply:

1. Ability to understand and comply with study procedures and give written informed consent
2. Following the diet and lifestyle recommendations at least 12 weeks prior to the treatment period
3. Males or post-menopausal females
4. Aged ≥18 years at the time of informed consent
5. Fasting serum TG levels ≥200 mg/dL (≥2.26 mmol/L) and ≤500 mg/dL (5.65 mmol/L) at screening
6. Serum HDL-C <50 mg/dL (<1.30 mmol/L) if male or <55 mg/dL (<1.42 mmol/L) if female at screening.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

1. Current or planned use of any lipid-altering medications other than the study drugs, statins, or ezetimibe during the study.

   i. Subjects currently on statins or ezetimibe must be at high risk for atherosclerotic CV diseases, and the dose(s) must be stable for at least 4 weeks prior to screening

   ii. For subjects currently on lipid-altering medications other than statins or ezetimibe, at least 4-week washout period (or for subjects currently on probucol at least 8 week washout period) will be required prior to the first fasting blood sampling at Screening Visit
2. Type 1 diabetes mellitus or poorly controlled Type 2 diabetes mellitus defined by HbA1c (NGSP level) ≥8.0% at screening
3. Uncontrolled hypertension defined by seated systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg at screening
4. Uncontrolled thyroid disorder
5. Creatinine ≥1.5 mg/dL at screening
6. Severe hepatic disorder defined as cirrhosis of Child-Pugh class B or C, or AST or ALT >2 × ULN at screening
7. History of pancreatitis
8. Gallbladder disorder, history of cholelithiasis, primary biliary cirrhosis, or history of disease or surgery that may affect the absorption, distribution, metabolism and excretion of drugs or the metabolism of bile salts
9. Unexplained creatine kinase (CK) >5 × ULN at screening
10. Myocardial infraction or stroke (including transient ischemic attack) within 3 months prior to the informed consent
11. New York Heart Association Class III or IV heart failure
12. History of malignancy within 5 years
13. Participation in another clinical study at the time of informed consent or administration of an investigational drug other than placebo within 16 weeks prior to the informed consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Percent change in fasting TG versus placebo from baseline to Weeks 8 and 12 | From baseline to Weeks 8 and 12
Percent change in fasting TG versus fenofibrate from baseline to Weeks 8 and 12 | From baseline to Weeks 8 and 12

SECONDARY OUTCOMES:
Percentage of patients who have achieved fasting TG <150 mg/dL at the end of the treatment period | At Week 12
Percent change from baseline to Weeks 8 and 12 in TC, LDL-C (direct method), LDL-C (Friedewald method), LDL-C (Martin/Hopkins equation), HDL-C (direct method), non-HDL-C (calculated), and remnant cholesterol (calculated) | From baseline to Weeks 8 and 12
Change from baseline to Weeks 8 and 12 in fasting TG, TC, LDL-C (direct method), LDL-C (Friedewald method), LDL-C (Martin/Hopkins equation), HDL-C (direct method), non-HDL-C (calculated), and remnant cholesterol (calculated) | From baseline to Weeks 8 and 12
Percent change from baseline to the end of the treatment period in Apo A1 and Apo B | From baseline to Week 12
Percent change from baseline to the end of the treatment period in TG/HDL-C, TC/HDL-C, non-HDL-C/HDL-C, LDL-C/HDL-C, LDL-C/Apo B, and Apo B/Apo A1 | From baseline to Week 12
The incidence of adverse events and adverse drug reactions after the administration of the study drug | Up to Week 12
Change from baseline to Week 4, 8, and 12 in clinical laboratory tests (chemistry, hematology), vital signs (BP [mmHg], PR [bpm], weight [kg], waist [cm], and BMI [kg/m^2]; each parameter is evaluated individually.), 12-lead ECGs | From baseline to Week 4, 8, and 12
Number and percentage of patients who experience laboratory abnormalities of special interest including, but not limited to ALT, AST, ALP, CK, and, creatinine during the treatment period | Up to Week 12

CONTACTS AND LOCATIONS:
Locations (33):
- China (33):
  - Huainan First People's Hospital, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Chengdu Xinhua Hospital, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fujian
  - Peking Union Medical College Hospital, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Guangxi
  - Hainan General Hospital, Hainan
  - The Second Hospital of Hebei Medical University, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Helongjiang
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology, Hubei
  - Tongji Hospital, Tongji Medical College of HUST, Hubei
  - Shaanxi Provincial People's Hospital, Hubei
  - The Third Xiangya Hospital of Central South University, Hunan
  - The Third Hospital of Changsha, Hunan
  - Nanjing Jiangning Hospital, Jiangsu
  - Sir Run Run Hospital Nanjing Medical Universtiy, Jiangsu
  - Affiliated Hospital of Jiangsu University, Jiangsu
  - Jiangxi Provincial People's Hospital, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Jiangxi
  - The First Hospital of Nanchang, Jiangxi
  - Jiu Jiang No. 1 People's Hospital, Jiangxi
  - Pingxiang People's Hospital, Jiangxi
  - China-Japan Union Hospital of Jilin University, Jilin
  - Shanghai Tongren Hospital, Shanghai
  - People's Hospital of Deyang City, Sichuan
  - Tianjin Union Medical Center, Tianjin
  - The Affiliated Hospital of Hangzhou Normal University, Zhejiang
  - People's Hospital of Wenzhou City, Zhejiang

REFERENCES:
- [Result] Dai W, Lv Q, Li Q, Fu L, Zhang Y, Zhang Y, Liu L, Tanigawa R, Kunitomi K, Kamei R, Suganami H, Ma C. Efficacy and Safety of Pemafibrate, a Novel Selective PPARalpha Modulator in Chinese Patients with Dyslipidemia: A Double-Masked, Randomized, Placebo- and Active-Controlled Comparison Trial. J Atheroscler Thromb. 2025 Feb 1;32(2):125-140. doi: 10.5551/jat.64112. Epub 2024 Aug 2. PMID 39098034